CLINICAL TRIAL: NCT00953329
Title: An Open-Label Study to Determine the Safety and Efficacy of Alefacept as Monotherapy in Subjects With Chronic Plaque Psoriasis Who Have Failed to Respond to Anti-TNF Therapy
Brief Title: Alefacept in Subjects With Chronic Plaque Psoriasis Who Failed to Respond to Anti-TNF Therapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Subjects declined enrollment; sponsor/PI elected to close study.
Sponsor: John Murray (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor-Investigator, John Murray, Professor of Dermatology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00002474; Funding Agency # ER-07-001; IND # 100770
Record Dates: First submitted 2009-07-22; First posted 2009-08-06 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Plaque Psoriasis
MeSH Terms: interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alefacept 15 mg IM qweek (Experimental): Alefacept will be given to subjects with plaque psoriasis who have failed treatment with Fnbrel.
  Interventions: Drug: alefacept

INTERVENTIONS:
Drug: alefacept — Alefacept 15 mg IM once a week were to be administered for 12 weeks, which is the FDA approved dosage, duration, and frequency. This study allowed an additional 8 doses if subject did not achieve a 'clear' response with the original 12 weeks of treatment. Each enrolled subject must have failed a response to anti-TNF therapy prior to entering this study.
  Other Names: Amevive

SUMMARY:
Study Status:

Duke University Health System Institutional Review Board has received notification of study termination; final IRB closure date is 12/12/2008. Study enrollment is now closed.

Enrollment Update:

Only one subject was entered into this study out of an expected enrollment of 15 patients in this single site clinical trial. With no recruitment interest, the financial sponsor and Sponsor-PI chose to close the clinical trial.

DETAILED DESCRIPTION:
This is an open-label study using alefacept in the treatment of patients with chronic plaque psoriasis who have not responded to treatment with an anti-TNF agent. Patients not responding to Enbrel® 50 mg weekly with a 75% reduction of Psoriasis Area and Severity Index (PASI) Score or a Physician Global Assessment (PGA) score of 'almost clear' or 'clear', will be treated with 15 mg alefacept intramuscularly (IM) once weekly for up to 20 weeks. Patients who have 'cleared' or 'almost cleared' at the end of 12 weeks of treatment with alefacept will have completed the 'standard treatment' phase of the study. Study subjects who have not responded to treatment during the initial 12 weeks will continue with alefacept therapy for an additional 8 weekly doses or until the subject has reached a PGA of 'almost clear' or 'clear'. Alefacept is FDA approved for this indication for 12 weeks of treatment and this clinical trial is extending the treatment window for up to 8 additional weeks. Because of this increased exposure to alefacept, all subjects will be carefully monitored while on treatment and followed post-treatment at 3, 4, 6, 9 and 12 months after the last dose of alefacept is given.

Purpose:

This open-label study will determine the safety and efficacy of Amevive® 15 mg IM weekly in subjects with chronic plaque psoriasis who have not sufficiently responded to etanercept, an anti-TNF agent. The plan also is to determine the length of response time to point of relapse and to determine the length of time before retreatment with alefacept is necessary.

Patient Population:

This study is for adult men and women, ages 18 to 80, with chronic plaque psoriasis. At the time of enrollment, the subject must have received 50 mg per week of Enbrel without achieving a response of 'almost clear' or 'clear' according to PGA or has not responded with a 75% reduction of PASI Score.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between ages of 18 and 80 years
* Subjects diagnosed with chronic plaque psoriasis who require systemic therapy.
* Must be receiving anti-TNF treatment without achieving response of 'almost clear' or 'clear' according to PGA or has not responded with 75% reduction PASI score.
* Must be willing to receive up to 20 weeks of IM injections weekly
* CD4 counts must be above 250 cells/mm3 at screening

Exclusion Criteria:

* Diagnosis of unstable erythroderma or pustular psoriasis or guttate psoriasis
* Serious local infection or systemic infection 3 months prior to receiving study drug.
* Subjects with CD4 lymphocyte count less than 250 cells/mm3 at study entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Murray, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment ended in Dec 2008. Clinical Trial was located in Medical Center Clinic.
Pre-assignment Details: No adverse events occurred
Period: Overall Study
Arm/Group | Alefacept Treated
Started | 1
Completed | 0
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Treatment Alefacept
Description: Terminated study
Time Frame: 12 weeks (study terminated)
Population: Study terminated
Groups:
- Alefacept: 50 mg
Arm/Group | Alefacept
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to one patient enrolled . The patient stopped the study because she was not improved and desired alternative treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No